CLINICAL TRIAL: NCT07123740
Title: Comparison of the Postoperative Analgesic Effects of Intrathecal Morphine and Bi-level Erector Spinae Plane Block in Liver Transplantation Donors
Brief Title: Comparison of the Postoperative Analgesic Effects of ITM and Bi-level ESPB in Liver Transplantation Donors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Atakan Sezgi, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-155
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Liver Transplantation; Pain Management
Keywords: Liver Transplantation; Intrathecal Morphine; Erector Spinae Plane Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Morphine (Active Comparator): An intrathecal injection of morphine 300μg will be administered at the L3-L4 or L4-L5 level.
  In the intraoperative period, intravenous meperidine 0.5 mg/kg will be given 30min before the end of surgery.
  Interventions: Procedure: Intrathecal Morphine
- Bi-level Erector Spinae Plane Block (Active Comparator): After the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T8 spinous process, 10 ml of 0.25% bupivacaine hydrochloride will be injected cauda-cranially into the interfacial space below the erector spinae muscle, above the transverse process. Next, the needle will be withdrawn till subcutaneously and the linear US probe will be placed 2-3 cm lateral to the T10 spinous process. Finally, 10 ml of 0.25% bupivacaine hydrochloride will be injected cranio-caudally into the interfacial space below the erector spinae muscle, above the transverse process.
  This procedure will be performed bilaterally. A total of 40 ml of 0.25% bupivacaine will be injected for bilateral and bi-level ESPB application.
  In the intraoperative period, intravenous meperidine 0.5 mg/kg will be given 30min before the end of surgery.
  Interventions: Procedure: Bi-level Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Intrathecal Morphine — An intrathecal injection of morphine 300μg will be administered at the L3-L4 or L4-L5 level.
  Additionally, in the postoperative period a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Intrathecal Morphine
Procedure: Bi-level Erector Spinae Plane Block — Bi-level erector spinae plane block will be performed on the patients using a total of 40 ml of 0.25% bupivacaine under ultrasound guidance.
  Additionally, in the postoperative period a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Bi-level Erector Spinae Plane Block

SUMMARY:
Liver transplantation is a life-saving procedure for patients with end-stage liver disease, and postoperative pain management is critical for optimizing donor recovery and overall outcomes. Poorly controlled pain following donor hepatectomy may reduce quality of life, delay mobilization, and contribute to the development of chronic pain syndromes.

Regional anesthesia techniques, such as intrathecal morphine and erector spinae plane block, have been utilized to enhance postoperative analgesia and reduce perioperative opioid requirements, potentially minimizing opioid-related adverse effects.

In this study, we aimed to compare the postoperative analgesic efficacy of intrathecal morphine and Bi-level erector spinae plane block in living liver donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* American Society of Anesthesiologists (ASA) score I-II
* Body Mass Index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Patients under 18 and over 65 years of age
* ASA score III and above
* Patients with a history of bleeding diathesis
* BMI below 18 or above 30 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | On the operation day
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 0st, 1st, 2nd,4th, 12th, and 24th hours after surgery.

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Intraoperative period
  Remifentanil consumption for intraoperative period will be recorded
Postoperative Opioid Consumption | On the operation day
  Opioid consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)